CLINICAL TRIAL: NCT03052166
Title: A Prospective Multi-center Case Collection Study of Breast Imaging Examinations From Women to Evaluate the Non-inferiority of QT Ultrasound Compared to Digital Mammography-Digital Breast Tomography (DM-DBT)
Brief Title: Case Collection Study to Determine the Accuracy, Call Back and Cancer Detection Rates of QT Ultrasound in Breast Imaging
Acronym: ACCRUE
Status: Completed | Type: Observational
Sponsor: QT Ultrasound LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BR005
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Breast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort A: The group of asymptomatic subjects who have been given BI-RADS 1 or 2 based on their most recent standard of care assessment. All subjects will receive a QT Ultrasound scan.
  Interventions: Device: QT Ultrasound scan
- Cohort B: The group of asymptomatic women who have been given BI-RADS categories 4 or 4a, 4b, 4c or 5 based on their most recent standard of care assessment. All subjects will receive a QT Ultrasound scan.
  Interventions: Device: QT Ultrasound scan
- Cohort C: The group of women who have been given BI-RADS categories 1, 2, 3, 4 or (4a, 4b, 4c), 5 or 6 based on their most recent standard of care assessment. All subjects will receive a QT Ultrasound scan. Subjects are assigned to Cohort C when it has been determined they cannot be assigned to Cohort A or Cohort B.
  Interventions: Device: QT Ultrasound scan

INTERVENTIONS:
Device: QT Ultrasound scan — QT Ultrasound scan

SUMMARY:
Brief Summary: The QT Ultrasound system is an automated scanner which transmits pulsed ultrasound plane waves through the breast, as well as collects reflected ultrasound output. As the patient lays prone on a table, the breast is submerged in a warm water bath. The transmitter and receiver assembly moves around the suspended breast to record data for successive sub-volumes of targeted tissue. More than 2000 elements in the curvilinear transducer's array encircle the breast to gather data from the tissue structures of the breast, from nipple to chest wall. Information gathered from this automated QT scan encompasses the entire breast which is currently not commercially available using any other ultrasound technology.

DETAILED DESCRIPTION:
This is a prospective, multicenter, multi-arm case collection study, with IRB approval. The study will follow an adaptive design with an initially planned total enrollment of approximately 600 cases to include both benign and malignant cases, representative of all tissue densities.

The images and clinical data accrued in this prospective case collection will be used for creation of a database to facilitate future reader's studies, publications, building teaching files, and future marketing for QT Ultrasound.

ELIGIBILITY:
INCLUSION CRITERIA All Subjects

1. Female
2. Age 18 or older
3. Willing to receive a QT Ultrasound Breast Scan
4. Willing and able to provide written Informed Consent prior to any research-related procedure(s)

Cohort A and B Subjects that do not meet these Inclusion Criteria will be evaluated for Inclusion in Cohort C

1. Eligible for routine screening mammography as per ACR guidelines
2. Willing and able to submit or complete at the clinical site a Digital Mammography with Digital Breast Tomosynthesis exam (to include Craniocaudal (CC) and Mediolateral Oblique (MLO) views - for one or both breasts, within 3 months, before or after, their QT scan.

Cohort C

1. Willing and able to submit available breast imaging - for one or both breasts, before or after, their QT scan.

EXCLUSION CRITERIA All Subjects

1. Pregnancy
2. Currently breastfeeding
3. Allergies to device materials
4. Physical inability to tolerate the procedure on the scanner, i.e. inability to lie prone and still for up to 30 minutes at a time
5. Open wounds, sores or skin rash present on the breast(s) or nipple discharge from the scanned breast
6. Breasts too large for scanner, i.e. inability to successfully "fit" breast after the subject is placed on scanner
7. Body weight greater than 400 lbs. (180 kg)
8. Has a concurrent disease or condition which in the judgment of the Principal Investigator disqualifies the subject, from participating in the study
9. Magnetic material in the chest which in the judgement of the Principal Investigator would interfere with or be impacted by the magnets within the study device.

Cohort A and B Subjects that meet any of these conditions below will not be eligible for Cohort A or B and will be evaluated for eligibility in Cohort C.

1. History of breast cancer in the past 12 months.
2. Most recent screening mammography exam was completed more than 3 months but less than 11 months prior.
3. History of breast surgeries or interventional breast procedures in the past 12 months, except for Fine Needle Aspiration(s) or Cyst Aspiration(s)

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women, age 18 and older
Sampling Method: Probability Sample
Enrollment: 755 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Comparison of QT Ultrasound to DM-DBT | 12 months
  Non-inferiority evaluation of sensitivity, specificity, positive predictive value and non-cancer recall rate.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Memorial Care Long Beach, Long Beach, California
  - Marin Breast Health Trial Center, Novato, California

IPD SHARING:
Plan to Share IPD: No